CLINICAL TRIAL: NCT06879691
Title: A Randomized Controlled Trial on the Efficacy and Pain Impact of Nimotuzumab Combined with a Painkiller in Comprehensive Treatment of Advanced Squamous Cell Carcinoma of Head and Neck
Brief Title: A Trial of Nimotuzumab and Pinkiller Efficacy and Pain in Advanced Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Collaborators: Baotou Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nimo-N&C-2021-03
Record Dates: First submitted 2025-02-24; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — nimotuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nimotuzumab group (Experimental): nimotuzumab, 200mg/w, for 6 weeks cis-platinum, 30mg/m2/w, for 6 weeks IMRT, 66～70Gy (2Gy/F, 35F), for 6 weeks painkiller, three ladders pain analgesic
  Interventions: Drug: Nimotuzumab; Drug: cis-platinum; Radiation: IMRT combine with cisplatin concurrent chemotherapy; Drug: painkiller
- control group (Other): cis-platinum, 30mg/m2/w, for 6 weeks IMRT, 66～70Gy (2Gy/F, 35F), for 6 weeks painkiller, three ladders pain analgesic
  Interventions: Drug: cis-platinum; Radiation: IMRT combine with cisplatin concurrent chemotherapy; Drug: painkiller

INTERVENTIONS:
Drug: Nimotuzumab — nimotuzumab group nimotuzumab, 200mg/w, for 6 weeks
  Other Names: H-R3
  Arms: nimotuzumab group
Drug: cis-platinum — 30mg/m2/w, for 6 weeks
  Other Names: cisplatin
Radiation: IMRT combine with cisplatin concurrent chemotherapy — IMRT, 66～70Gy (2Gy/F, 35F), for 6 weeks
Drug: painkiller — three ladders pain analgesic( First step: For mild pain, non-opioid agents (excluding nonsteroidal anti-inflammatory drugs [NSAIDs]) combined with adjuvant analgesics are administered; Second step: For moderate pain, weak opioids combined with NSAIDs and adjuvant analgesics are prescribed;Third step: For severe pain, strong opioids combined with NSAIDs and adjuvant analgesics are used.)

SUMMARY:
The purpose of this study is to investigate the impact of combining Nimotuzumab with analgesic agents on pain management outcomes, as well as the effectiveness and safety profile of this therapeutic combination in the comprehensive treatment of locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
The study is an open-label, randomized controlled phase II clinical trial designed to evaluate the impact of Nimotuzumab combined with analgesic therapy on pain management outcomes, as well as the therapeutic efficacy and safety profile of this combination in the comprehensive treatment of locally advanced head and neck squamous cell carcinoma.

Eligible participants will be randomly assigned to either the experimental group or the control group. Patients in the experimental group will receive Nimotuzumab plus analgesic therapy in addition to concurrent radiochemotherapy, while those in the control group will undergo analgesic therapy combined with concurrent radiochemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, inclusive of 18 years but exclusive of 75 years.
* ECOG Performance Status (PS) score 0-2.
* Histologically or cytologically confirmed Stage III-IVb (according to the 2020 CSCO Guidelines for Diagnosis and Treatment of Head and Neck Tumors) squamous cell carcinoma of the head and neck (including oral, oropharyngeal, hypopharyngeal, and laryngeal cancers; excluding nasopharyngeal carcinoma).
* EGFR-positive expression confirmed by immunohistochemistry.
* Patients deemed ineligible for surgery (due to physical contraindications or refusal of surgery).
* At least one measurable lesion according to RECIST 1.1 criteria:

CT scan ≥10 mm (tumors not measurable by calipers should be recorded as non-measurable).

Chest X-ray ≥20 mm. Pathologically enlarged lymph nodes: short-axis ≥15 mm on CT scan (slice thickness ≤5 mm).

Suitable for comprehensive treatment with curative or palliative intent. ●Baseline pain assessment: Numeric Rating Scale (NRS) score ≥1. Patients not previously treated with opioids who are candidates for opioid therapy.

Patients on weak opioids with inadequate pain control requiring escalation to strong opioids.

Patients with moderate-to-severe cancer pain on strong opioids with inadequate control.

Patients requiring urgent intervention due to poorly controlled pain.

* Expected survival ≥3 months.
* Adequate hematologic function:

White blood cell count ≥4×10^9/L. Absolute neutrophil count ≥1.5×10^9/L. Platelets ≥100×10^9/L. Hemoglobin ≥90 g/L.

●Adequate renal function: Serum creatinine ≤1.2 mg/dL or creatinine clearance ≥60 mL/min.

●Adequate hepatic function: Total bilirubin ≤1.5×ULN (≤3.0×ULN if liver metastases present). AST and ALT ≤2.5×ULN (≤5.0×ULN if liver metastases present).

* Negative urine pregnancy test for female patients of childbearing potential (excludes those with bilateral oophorectomy, hysterectomy, or postmenopausal status).
* Signed informed consent.

Exclusion Criteria

* Received radiotherapy, chemotherapy, monoclonal antibody therapy, oral EGFR-TKI therapy, anti-angiogenic agents, or immunosuppressants within the past 6 months.
* Participation in another interventional clinical trial within 30 days prior to screening.
* Presence of distant metastases.
* History of other malignancies (except cured cervical carcinoma in situ, basal cell carcinoma of the skin, or malignancies cured ≥5 years prior).
* Uncontrolled comorbidities (e.g., heart failure, diabetes, hypertension, thyroid disorders, psychiatric diseases).
* Active HIV infection, viral hepatitis, or severe active infections (>Grade 2 per CTCAE v5.0).
* Chronic steroid therapy (>10 mg/day prednisone equivalent for >6 months).
* Known hypersensitivity to any component of the study drugs.

  ●≥Grade 2 peripheral neuropathy or hearing loss (per NCI CTCAE v5.0).
* Pregnancy, lactation, or refusal to use effective contraception (for both male and female participants) until 6 months after the last treatment.
* Investigator judgment of unsuitability for the study.
* Unwillingness or inability to provide informed consent.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by INV per RECIST v1.1.cause,whichever occurs first.

SECONDARY OUTCOMES:
NRS score | Baseline, during concurrent radiochemotherapy (weeks 1,6), post-intervention (week 7), every 3 months for first 2 years, then every 6 months thereafter (through study completion, average 4 years).
  NRS score, also known as numerical scoring method, is a commonly used method for assessing pain levels. It uses a straight line or scale to allow patients to choose a number based on their personal pain perception, ranging from 0 (painless) to 10 (most painful) to indicate the degree of pain.
OS | From randomization to death from any cause (up to approximately 36 months)
  Refers to the time from randomization to death caused by any reason.

CONTACTS AND LOCATIONS:
Overall Officials: BO HAN, Study Director — Baotou Cancer Hospital
Locations (1):
- Baotou Cancer Hospital, Baotou, Inner Mongolia, China